CLINICAL TRIAL: NCT02082886
Title: Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) For Peritoneal Surface Malignancies Including Carcinomatosis or Sarcomatosis - Data Registry
Brief Title: HIPEC For Peritoneal Surface Malignancies Including Carcinomatosis or Sarcomatosis - Data Registry
Status: Completed | Type: Observational
Sponsor: Edward-Elmhurst Health System (Other)
Responsible Party: Sponsor
Other Study IDs: EDW120613A
Record Dates: First submitted 2014-03-05; First posted 2014-03-10 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Peritoneal Neoplasms; Neoplasm Metastasis; Adenocarcinoma; Sarcoma
Keywords: Metastasis; Carcinomatosis; Carcinosis; Sarcomatosis; CRS; Cytoreductive surgery; HIPEC; Heated Intraperitoneal Chemotherapy; Intra-abdominal; Sugarbaker technique; Mitomycin C; Cisplatin; Doxorubicin; Oxaliplatin; Melphalan
MeSH Terms: conditions — Peritoneal Neoplasms; Neoplasm Metastasis; Adenocarcinoma; Sarcoma; Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
In this registry study the investigators will collect data about patients' disease, treatment, and response to treatment to include in both our local and national databases. These can then be used by investigators to answer questions about cytoreductive surgery/HIPEC such as how well-tolerated or effective it is in specific populations.

DETAILED DESCRIPTION:
Patient Selection: The sole inclusion criteria for this study will be those consenting patients who are to undergo cytoreductive surgery followed by HIPEC.

Data Collection and Use Plan: For those patients who provide informed consent, data listed below will be collected during and after treatment. This will be entered into the PI's local database for future use and, after being de-identified, will be shared with a national database (held by the American Society of Peritoneal Surface Malignancies) to bolster the amount available for researchers looking at efficacy and outcomes such as overall survival rates, progression-free survival, and tolerability in certain populations.

Data Collected (as applicable): Age, primary tumor, dates of prior surgeries, prior chemotherapy with dates and whether it was neoadjuvant in nature, length of disease status, comorbidities, Peritoneal Surface Disease Severity Score, Peritoneal Cancer Index as determined prior to surgery, Peritoneal Cancer Index as determined during surgery, Completeness of Cytoreduction score, ascites present, blood products used, complications, length of stay in ICU and in hospital, where discharged, death within 30 days, readmission and reason, date of recurrence, treatment of recurrence, and time from procedure to death. For the HIPEC surgical procedure itself, data collected will be: date, duration, chemotherapeutic used and dose, duration of circulation, fluid temp, and flow rate.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to undergo cytoreductive surgery followed by HIPEC performed by the PI at Edward Hospital
* Provides consent by signing informed consent form

Exclusion Criteria:

* Not eligible for surgery or for potential cytoreductive surgery and/or HIPEC as determined by the PI
* Does not consent to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sole inclusion criteria for this study will be those consenting patients who are to undergo cytoreductive surgery followed by HIPEC performed by the PI at Edward Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2014-02; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | From time of treatment until death, approximately 10 years
  Collect data from patients undergoing CRS/HIPEC which will be used to examine overall survival rates in specific patient populations.

SECONDARY OUTCOMES:
Progression-free survival rate | From time of treatment until time of disease progression, approximately 10 years
  Collect data from patients undergoing CRS/HIPEC which will be used to examine progression-free survival rates in specific patient populations
Rates of complications | During procedure until approximately 90 days post
  Collect data from patients to examine rates of complications in specific patient populations

CONTACTS AND LOCATIONS:
Overall Officials: George I Salti, MD, Principal Investigator — Edward-Elmhurst Healthcare
Locations (2):
- United States (2):
  - Elmhurst Memorial Health Care, Elmhurst, Illinois
  - Edward Hospital, Naperville, Illinois

REFERENCES:
- See also: Related Info — http://www.edward.org/cancersurgery